CLINICAL TRIAL: NCT06716034
Title: Mood And Kids diEt (MAKE-It): A Pilot Randomized Controlled Trial for a Personalized Dietary Intervention for Adolescents With Depression
Brief Title: Mood And Kids diEt (MAKE-It) Pilot Trial
Acronym: MAKE-IT pRCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Daphne Korczak, Associate Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MAKE-IT pRCT
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-10

CONDITIONS: Depression - Major Depressive Disorder; Adolescent
Keywords: adolescent; diet; depression; randomized controlled trial; pilot
MeSH Terms: conditions — Depression | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized Nutrition Plan and Support (Experimental): This group will receive the nutrition intervention
  Interventions: Other: Personalized Nutrition Plan and Support
- Control (No Intervention): This group will receive information about Canada's food guide, a recommended healthy diet.

INTERVENTIONS:
Other: Personalized Nutrition Plan and Support — The intervention is a virtually-delivered, personalized nutrition plan and support to improve dietary intake of healthy food (fruit, vegetables and whole grains), based on the principles of a Mediterranean-style diet. Components of the intervention include nutrition counselling, menu planning and the provision of groceries, delivered biweekly, face-to-face, by a registered dietitian over 8 weeks, using a virtual platform. The nutrition counselling structure is grounded in evidence-based behaviour change theory for dietary interventions. Youth and parents will co-develop a personalized menu plan. In addition to biweekly nutrition counselling, participants will receive a food pantry basket, and weekly grocery deliveries to support the menu plan.
  Arms: Personalized Nutrition Plan and Support

SUMMARY:
This study is being done to examine the feasibility, including recruitment, retention and acceptability of a randomized controlled trial of a personalized dietary intervention in adolescents with depression. Evidence suggests that dietary quality may affect an individual's mood. A healthy diet includes vegetables, fruit, nuts, seeds, and olive oil, as well as minimally processed whole grains, legumes, and moderate amounts of lean meat, fish, and dairy.

The investigators will examine the feasibility of testing a personalized nutrition eating plan in a study that uses a randomized controlled trial design for children and youth with depression.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MDD
* Center for Epidemiological Studies Depression Scale for Children (CESD-C) score ≥ 25 at baseline
* access to the internet and a computer or smart phone
* presence of a parent who is willing to participate

Exclusion Criteria:

* adherent to a high-quality diet at baseline
* presence of an eating disorder
* currently participating in other dietary programs or studies
* actively attempting to increase or decrease body weight;
* presence of a chronic medical condition;
* unstable psychiatric condition (e.g., mania, active suicidal ideation)

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Intervention | Baseline, 9 weeks
  Feasibility of Intervention Measure (FIM). The FIM is a self-reported four-item measure scored using a five-point Likert scale ranging from 'completely disagree' (1) to 'completely agree' (5) with higher scores indicating greater acceptability or feasibility. Higher scores indicate greater feasibility with a maximum score of 20. Parents and youth will complete this measure.
Acceptability of the Intervention | Baseline, 9 weeks
  Acceptability of Intervention Measure (AIM). The AIM is a self-reported four-item measure scored using a five-point Likert scale ranging from 'completely disagree' (1) to 'completely agree' (5) with higher scores indicating greater acceptability or feasibility. Higher scores indicate greater acceptability with a maximum score of 20. Parents and youth will complete this measure.

SECONDARY OUTCOMES:
Depression Symptoms | Baseline, 9 weeks
  Self-reported depression severity will be measured using the Centre for Epidemiological Studies Depression - Children (CES-DC) instrument, a 20 item youth-report measure that assesses symptoms of depression with demonstrated good reliability and validity. Participants will be asked to rate their depression symptoms on a 4-point Likert scale. Higher scores represent greater symptom severity with a maximum potential total score of 60. Youth will complete this measure.
Depression Symptoms | Baseline, 9 weeks
  Clinician-rated depression symptoms will be assessed using the Children's Depression Rating Scale Revised (CDRS-R). The CDRS-R, a semi-structured clinical interview which takes 15-20 min to administer, is a widely used interviewer-administered rating scales for measuring depression symptoms in intervention studies of adolescent depression. The measure assesses depression symptoms, rated on 5- to 7-point Likert rating scales. Depression symptom domains are aligned with the diagnostic criteria for depression and include sleep disturbance, excessive fatigue, suicidal ideation, and social withdrawal. Participants are asked about information on 14 items. Youth will complete this measure.
KIDMED2 | Baseline, 9 weeks
  The 'KIDMED2' questionnaire will evaluate dietary intake in relation to the Mediterranean Diet in children and adolescents. KIDMED2 is a 16-item questionnaire that can be self-administered or conducted by an interview with responses being yes/no. Items related to lower adherence are assigned a value of -1 (4 items) and those related to higher adherence +1 (12 items). Scores range from 0-12. A total score of ≤ 3 is considered poor adherence; a score of 4-7 is considered medium adherence and ≥8 is high adherence. Youth will complete this measure.
Automated Self-Administered 24-Hour (ASA24) Dietary Assessment | Baseline, 9 weeks
  The National Cancer Institute's Automated Self-Administered 24-Hour (ASA24) Dietary Assessment is a validated tool that employs the Automated Multiple-Pass Method and is freely available in the public domain. Usual or habitual dietary intake requires two ASA24 dietary intake measures one during the week and another on a weekend day. Reported energy intake (rEI) and nutrient intakes will be generated automatically by the ASA24 software using the ASA24-Canada-2018 version, released in April 2019 and food composition data from the Canadian Nutrient File as well as data from the Food and Nutrient Database for Dietary Studies. Youth will complete this measure.
Food Choice Questionnaire | Baseline, 9 weeks
  The Food Choice Questionnaire is a 36-item self-administered questionnaire that evaluates factors which influence dietary choices. Factors which might influence food choices are divided into 9 subscales, which are labelled health, mood, convenience, sensory appeal, natural content, price, weight control, familiarity and ethical concern. Items are scored on a 4-point Likert scale ranging from 1 (not important at all) to 4 (very important). Higher subscale scores reflect a greater emphasis on that particular factor when selecting foods. Youth will complete this measure.
Diet Satisfaction | Baseline, 9 weeks
  Diet satisfaction will be assessed using the Diet Satisfaction Score (DSS), a comprehensive tool consisting of 10 items focused on measuring a singular dimension. The DSS demonstrates strong reliability through a robust intraclass correlation coefficient of 0.64. Moreover, the minimal mean difference (95% confidence interval, CI) between repeated test scores stands at 0.03 (-0.02, 0.09), affirming its stability. Participants rate their level of agreement on a 5-point Likert-type scale across the 10 statements, spanning from 'strongly agree' to 'strongly disagree.' Higher scores on this scale directly correlate with greater satisfaction with the diet. Calculated as the mean of all items, the total score ranges from 1 to 5, with 5 signifying optimal satisfaction. Higher scores indicate a stronger sense of satisfaction with the diet. Youth will complete this measure.
International Physical Activity Questionnaire for Adolescents (IPAQ-A) | Baseline, 9 weeks
  The International Physical Activity Questionnaire for Adolescents (IPAQ-A) is a self-reported questionnaire that measures physical activity (PA) in the last 7 days. Participants will estimate the number of occasions per week for activities such as sitting, walking, leisure cycling, running and/or aerobics. The total number of days and minutes of PA will be reported as metabolic equivalent of task (MET) per hour per week, with greater METs indicating greater physical activity. Using the IPAQ scoring protocol, PA will be reported as a continuous variable - the metabolic equivalent of task (MET) minutes per week and as a three-level categorical variable (using IPAQ-A cut-points): low level of activity; moderate level of activity; or high level of activity. Youth will complete this measure.
Dutch Eating Behavior Questionnaire | Baseline, 9 weeks
  Eating behaviour will be assessed with The Dutch Eating Behavior Questionnaire (DEBQ), a 33-item self-report questionnaire to comprises three scales assessing restrained eating (DEBQ-R), emotional eating (DEBQ-E), and external eating (DEBQ-X) behaviour. Items on the DEBQ range from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behaviour. A score of 15 or higher indicates a risk for depression in children and adolescents. The scale has demonstrated good to excellent internal consistency (α = 0.84 - 0.92) and factorial validity. Youth will complete this measure.
Pittsburg Sleep Quality Index (PSQI) | Baseline, 9 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-reported questionnaire designed to assess sleep quality and disturbances within a one-month timeframe. It comprises 19 individual items contributing to the calculation of seven "component" scores each scored 0 (no difficulty) to 3 (severe difficulty): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of these seven component scores yields one global score ranging from 0 to 21 with the higher total score indicating worse sleep quality. In distinguishing between good and poor sleepers, a global PSQI score > 5 yields a sensitivity of 89.6% and a specificity of 86.5%. Youth will complete this measure.
Parent Food Modelling | Baseline, 9 weeks
  Parental food modelling is evaluated with 10 items adapted from Cullen's scale, each rated on a four-point Likert scale from 'Never' (0) to 'Always' (3) which has been used to predict diet outcomes in adolescent samples. Higher scores signify greater healthful parental food modeling, with a maximum score of 30. Youth will complete this measure.
Satisfaction with menu planning | Baseline, 9 weeks
  Satisfaction with menu planning is evaluated through a single item, independently assessed by parents and adolescents using a five-point Likert scale that ranges from 'very dissatisfied' (1) to 'very satisfied' (5). Parents and youth will complete this measure.
Satisfaction with nutrition counselling sessions | Baseline, 9 weeks
  Satisfaction with nutrition counseling sessions is evaluated through a single item, independently assessed by parents and adolescents using a five-point Likert scale that ranges from 'very dissatisfied' (1) to 'very satisfied' (5). Parents and youth will complete this measure.
Nutrition Attitude and Knowledge Questionnaire | Baseline, 9 weeks
  The Nutrition Attitudes and Knowledge (NAK) questionnaire is a brief questionnaire developed by a team of educators and dietitians to assess knowledge of the 2019 Canada Food Guide. We have adapted the NAK for this study. The adapted NAK questionnaire contains 22 items, with one section evaluating nutrition attitudes and four sections assessing nutrition knowledge associated with the different food groups. The nutrition attitudes section contains four 5-point Likert scale questions (e.g., "Eating healthy now can help me be healthy in the future"), with higher scores indicating more positive attitudes about nutrition. Thirteen multiple choice and five true/false questions were developed to reflect knowledge of the CFG food groups: Drinks, Whole Grain Foods, Vegetables and Fruit, and Protein foods (both animal and plant-based). Parents and youth will complete this measure.
Screen time Questionnaire | Baseline, 9 weeks
  The Questionnaire for Screen Time of Adolescents (QueST) is a self-reported questionnaire to assess screen time on a typical day. Participants are asked how much time they spend on screens across five constructs: studying, working/internship-related activities, watching videos, playing games, and using social media/chat applications on weekdays and again on weekends. Items are summed to obtain total weekday and weekend screen time. The QueST test-retest intra-class correlation coefficients range from 0.76 for social media use on weekdays to 0.24 for watching videos on weekends. Youth will complete this measure.
Family and Nutrition and Physical Activity | Baseline, 9 weeks
  The Family and Nutrition and Physical Activity (FNPA) screening tool is a behaviorally-based assessment designed to allow parents to evaluate the family food environment and practices. FNPA has been extensively used in child and adolescent obesity research but also in studies examining diabetes prevention, family eating behaviour and cardiovascular risk factors.
  The FNPA is a 20-item screening tool with 10-constructs. Parents are asked to rate their child's behaviour on a 4-point Likert scale ranging from almost never to very often. 6 items are reverse scored for the following questions and construct 3-Family Eating Practices, 4- Family Eating Practices, 5-Food Choices, 7-Beverage Choices, 10-Restriction/Reward, 13-Healthy Environment. Higher scores reflect more healthy home environments since no cut points or thresholds have been established for determining healthy vs unhealthy home environments. Parents will complete this measure.
Screen for Child Anxiety Related Disorders | Baseline, 9 weeks
  Screen for Child Anxiety Related Disorders (SCARED) and the Revised Children's Anxiety and Depression Scale (RCAD) contains 41 items and measures rated on 3-point Likert-type scale anxiety using four domains: panic/somatic, separation anxiety, generalized anxiety, and school phobia with three possible responses ranging from ' not true or hardly ever true' to very often true or often true'. Parents will complete this measure.
The Revised Child Anxiety and Depression Scale (RCADS) | Baseline, 9 weeks
  The Revised Child Anxiety and Depression Scale - Parent Version (RCADS-P) is a 47-item self-report questionnaire with subscales including separation anxiety disorder (SAD), social phobia (SP), generalized anxiety disorder (GAD), panic disorder (PD), obsessive-compulsive disorder (OCD), and major depressive disorder (MDD). It also yields a Total Anxiety Scale (sum of the 5 anxiety subscales) and a Total Internalizing Scale (sum of all 6 subscales). Items are rated on a 4-point Likert scale from 0 ("never") to 3 ("always"). Parents will complete this measure.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No